CLINICAL TRIAL: NCT06756100
Title: Composition and Metabolic Activity of Gut Microbiota to Predict Early Inflammatory Bowel Disease Progression
Brief Title: Early Inflammatory Bowel Disease Progression
Acronym: PRO-IBD
Status: Recruiting | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Fondo Nacional de Desarrollo CientÃ-fico y TecnolÃ³gico, FONDECYT (Chile). (Unknown)
Responsible Party: Principal Investigator, Cristian Hernández Rocha, Academic, Pontificia Universidad Catolica de Chile
Other Study IDs: 1230757
Record Dates: First submitted 2024-09-30; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease (CD); Ulcerative Colitis (UC)
Keywords: Inflammatory bowel disease; Microbiome; Prediction
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Blood (DNA and serum), stool and biopsy samples (obtained during colonoscopy). Mucosal-luminal interface samples (Mucosal lavage samples)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IBD: Patients with gastrointestinal symptoms for at least 3 weeks suggesting IBD in whom IBD is confirmed
- Controls: Patients with gastrointestinal symptoms for at least 3 weeks suggesting IBD in whom IBD is ruled-out

SUMMARY:
The purpose of this study is to assess the capacity of the gut microbial composition and function to predict the course of IBD during the first year after diagnosis.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD), comprising Crohn ́s disease (CD) and ulcerative colitis (UC), is an idiopathic inflammatory condition of the gastrointestinal tract which is characterized by alternating periods of active disease and remission. IBD is often progressive and associated with significant morbidity. A common endpoint for a progressive course of CD or UC is the need for treatment escalation; initially with immunomodulators and subsequently - if disease activity persists - with biologic therapy or surgery. Early use of biologic therapy improves clinical outcomes and can prevent complications such as strictures, fistulae or severe and progressive disease, obviating need for surgery. The success of early initiation of biologic therapy is most likely related to a therapeutic "window of opportunity" for the implementation of effective therapies in patients with rapidly progressive disease. However, indiscriminate use of biologic therapy would entail exposure of IBD patients with indolent disease to unnecessary expensive treatments and their associated side effects. Unfortunately, the need for biomarkers to reliably guide IBD treatment in a timely manner remains unmet. The literature supports a relevant role for host-gut microbiota interactions in IBD progression. This interaction is often mediated by microbial-derived metabolites. Fecal short chain fatty acids (SCFA) and secondary bile acids (BA) are remarkable examples of such metabolites. They are reduced in IBD patients, and in animal models are capable of mitigating exaggerated host immune response with consequent improvement in gut inflammation. Recently, researchers have started to explore the capacity of taxonomic and metabolomic signatures to predict meaningful clinical outcomes in IBD. Given the role of gut microbes and their metabolites in immune response, they are plausible biomarkers of IBD progression and therapy response. However, most of the studies exploring biomarkers for IBD include patients with longstanding IBD or previous failure to first-line therapies, rendering their results incompatible with early risk stratification. An inception cohort of newly diagnosed IBD patients integrating clinical, transcriptomics, microbial and metabolomic profiling can overcome these limitations, increasing the sensitivity to detect biomarkers of progressive disease before the therapeutic "window of opportunity" has passed. In the clinical setting, such biomarkers would enable clinicians to maximize therapeutic efficacy of biologic agents and implement as early as IBD diagnosis, a cost-effective therapeutic approach.

The objective of this project is to establish whether an impaired gut microbial capacity to synthesize SCFA and secondary BA at the time of IBD diagnosis can predict early need for treatment escalation (progression). To achieve this objective, our specific aims are:

1) To define the gut taxonomic and metabolomic profiles of newly diagnosed IBD patients and their associations with early clinical outcomes. The investigators will recruit an inception cohort of treatment-naïve IBD patients before undergoing their first diagnostic colonoscopy. The global metabolome, including SCFA and secondary BA abundance will be analyzed, as well as the taxonomic profile of fecal samples and mucosal-luminal interface (MLI) aspirates obtained at colonoscopy. The identified "omics" signatures will be correlated to the need for treatment escalation to derive predictive biomarkers of progressive IBD course. 2) To establish the impact of gut microbial dysbiosis and dysmetabolism of SCFA and BA of newly diagnosed IBD patients on mucosal inflammation and host gene expression. Analysis of taxonomic and metabolomics profiles obtained in MLI samples will be integrated to mucosal host gene expression analysis to identify host transcripts affected by differential SCFA and secondary BA abundance.

3) To quantify the in vitro capacity of gut microbiota of newly diagnosed IBD patients to synthesize SCFA and secondary BA. Gut microbiota from IBD patients will be inoculated into a batch bioreactor which closely mimics the gut luminal environment. The investigators will then perform serial measurements of SCFA, BA and bacterial abundance, estimating rates of metabolite synthesis. The metabolic activity will be correlated to in vivo metabolite abundance and clinical outcomes.

The investigators anticipate that IBD patients requiring early therapy escalation (progressors) will have decreased in vivo concentrations of SCFA and secondary BA, and an impaired in vitro microbial capacity to synthesize these compounds compared to patients not requiring therapy escalation. The investigators also expect to find that the taxonomic and metabolomic signatures of these patients have a distinct impact on host gene expression. Our comprehensive approach will allow us to identify reliable biomarkers which can be exploited in the clinical setting to guide early biologic treatment using a 'personalized medicine' approach and will provide novel insight into the biologic mechanisms underlying need for premature therapy escalation as a proxy of early progressive and aggressive course in IBD.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with with at least 3 weeks of gastrointestinal symptoms including diarrhea, rectal bleeding, abdominal pain, tenesmus or urgency

Exclusion Criteria:

* Confirmed infectious disease of the gastrointestinal tract

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients attending the gastroenterology clinic at Pontificia Universidad Católica of Chile with at least 3 weeks of GI symptoms including diarrhea, rectal bleeding, abdominal pain, tenesmus or urgency will be identified by members of the Gastroenterology Medical Group. As part of standard of care (SOC), these patients will undergo stool testing to rule out gastrointestinal infections followed by full colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Compare gut microbiome composition and function from different sample types among participants with gastrointestinal symptoms with and without confirmed IBD by colonoscopy and biopsy | 36 months
  Researchers will obtain stool (before diagnostic colonoscopy), biopsy specimens (frozen and RNAlater stored samples), and intestinal washing (mucosal-luminal interface samples at colonoscopy)
In patients with confirmed IBD, researchers will identify whether there are differences in gut microbiome composition and function between patients who need therapy escalation (progressors) within the first 12 months after diagnosis | 12 months
  IBD patients who need therapy escalation (progressors) will be those who:
  * Undergo surgery (colectomy or small bowel resection) within the first year after diagnosis
  * Start biologic therapy within the first year after diagnosis
  * Do not achieve clinical remission at week 24 (Average daily stool frequency (SF) ≤1.5 and abdominal pain (AP) score ≤1.0 for Crohn's disease (CD), and rectal bleeding (RB) = 0 and SF score <2 on the patient reported outcome measure (PROM) component of the Mayo score for ulcerative colitis (UC) and IBD-unclassified (IBD-U).
  * IBD patients with fecal calprotectine ≥250 mcg/g at week 24

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Hernández-Rocha, MD, Principal Investigator — Pontificia Universidad Catolica of chile
Locations (1):
- Pontificia Universidad Catolica of Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided